CLINICAL TRIAL: NCT06638307
Title: A Phase 1, First-in-Human Study of MEN2312, a KAT6 Inhibitor, as Monotherapy and in Combination in Participants With Advanced Breast Cancer
Brief Title: A First-in-Human Study of MEN2312 in Adults With Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEN2312-01; 2024-514661-19-00 (EU CTIS Number); U1111-1308-5349 (Other: UTN number)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Cancer
Keywords: First-In-Human; MEN2312; Advanced Breast Cancer; KAT6
MeSH Terms: interventions — elacestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEN2312: Monotherapy (Experimental): Participants will receive MEN2312.
  Interventions: Drug: MEN2312
- MEN2312: Combination Therapy (Elacestrant) (Experimental): Participants will receive MEN2312 in combination with elacestrant.
  Interventions: Drug: MEN2312; Drug: Elacestrant

INTERVENTIONS:
Drug: MEN2312 — MEN2312 administered as oral tablets.
Drug: Elacestrant — Elacestrant administered as oral tablets.
  Other Names: Orserdu
  Arms: MEN2312: Combination Therapy (Elacestrant)

SUMMARY:
This is a first-in-human study of MEN2312, a lysine acetyltransferase 6 (KAT6) inhibitor, in adult participants with advanced breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy.
* Participant must have received at least one prior line of endocrine therapy for advanced/metastatic disease or participant who has radiological evidence of breast cancer recurrence or progression during or within 12 months from the end of or during adjuvant treatment with endocrine therapy, as these participants are considered as first-line relapsed participants. Progression on previous cyclin-dependent kinase 4/6 inhibitor treatment in combination with fulvestrant or aromatase inhibitor is required. No other therapeutic options are considered appropriate by the investigator.
* Up to 6 prior lines of systemic therapy (including up to 2 prior lines consisting of chemotherapy, cytotoxic antibody drug conjugate, or a combination of both regimens) are allowed in the advanced/metastatic setting.
* Presence of genetic alterations in PIK3CA/AKT1/PTEN in participants' tumor tissue.

Key Exclusion Criteria:

* Active or newly diagnosed central nervous system metastases.
* Participants with advanced, symptomatic visceral spread, who are at risk of life-threatening complications in the short term, including massive uncontrolled effusions (peritoneal, pleural, pericardial), pulmonary lymphangitis, or liver involvement >50%.

Note: Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting Toxicity When Administered MEN2312 | Baseline through Day 28
Recommended Phase 2 Dose (RP2D) of MEN2312 | Baseline through Month 6

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Baseline through 28 days after the last treatment administration (up to approximately 7 months)
Duration of Response (DOR) | Baseline through 28 days after the last treatment administration (up to approximately 7 months)
Clinical Benefit Rate (CBR) | Baseline through 28 days after the last treatment administration (up to approximately 7 months)
Progression-free Survival (PFS) | Baseline through 28 days after the last treatment administration (up to approximately 7 months)
Overall Survival (OS) | Baseline through 3 months after the last treatment administration (up to approximately 9 months)
Time to Response (TTR) | Baseline through 28 days after the last treatment administration (up to approximately 7 months)
Area Under the Plasma Concentration-time Curve (AUC) of MEN2312 When Administered as Monotherapy | Up to 6 months post dose
AUC of MEN2312 When Administered as Combination Therapy | Up to 6 months post dose
Amount of MEN2312 Excreted in Urine When Administered as Monotherapy | Up to 2 months post dose
Comparison of Plasma Concentration of MEN2312 Monotherapy With MEN2312 Combination Therapy | Up to 6 months post dose

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Highlands Oncology Group, Springdale, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Hematology Oncology - Parkside, Santa Monica, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Advent Health Orlando, Altamonte Springs, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists & Research Institute (FCS) - Sarasota, Sarasota, Florida
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - START Midwest - Oncology, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Astera Cancer Care, East Brunswick, New Jersey
  - SCRI Oncology Partners Group, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - START San Antonio, LLC, San Antonio, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - START Mountain, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia